CLINICAL TRIAL: NCT02020473
Title: Informed Consents for Withholding/Withdrawing Life Support in Intensive Care Units
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2012-0858
Record Dates: First submitted 2013-12-12; First posted 2013-12-25 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-12

CONDITIONS: Death Occurring in Intensive Care Units
Keywords: Informed consents; Withholding/withdrawing life support (WLS); Intensive care unit (ICU)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- WLS group: patients with informed consents for withholding/withdrawing life support
- non-WLS group: patients without informed consents for withholding/withdrawing life support

SUMMARY:
End-of- life care is a major issue in medical ethics with life support technology progress. Intensive care may prolong the dying process in patients who have been unresponsive to the treatment already provided. Withholding or withdrawing of life support (WLS) care was introduced to avoid the suffering of critically ill patients. Decision to WLS is a difficult and affected by several factors including not only disease severity but also ethics, religion, culture, and legal background. In western countries, advance directives had an important role to WLS for dying patients and honor patient autonomy. However, the illegality of advance directives in Korea and Korean culture under Confucianism, requiring children to do the best to treat their parents in the name of filial piety make physicians and family members difficult to WLS in terminally ill patients.

Additionally, WLS in intensive care unit had been usually decided without official documentation before the final legal decision by Supreme Court in Korea. Scanty information exists about end-of-life practices because informed consents of WLS were taken after the legal decision.

Thus, we aimed to investigate the current status of informed consent at the time of decision to WLS and difference between WLS group and non-WLS group in Korea.

ELIGIBILITY:
Inclusion Criteria:

* patients who died from January 2012 to December 2012 in the surgical or medical Intensive Care Unit (ICU) at Severance Hospital, Yonsei University Health System, in Seoul, Korea.

Exclusion Criteria:

* Patients diagnosed with brain death

Max Age: 92 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who died from January 2012 to December 2012 in the surgical or medical Intensive Care Unit (ICU)
Sampling Method: Non-Probability Sample
Enrollment: 348 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Signing of informed consents for withholding/withdrawing life support | 1 year after ICU admission
  Primary outcome was existence of informed consents for withholding/withdrawing life support. Data from informed consents for WLS included main family members who signed the WLS and type of the life support modalities withheld or withdrawn.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Chief of ICUs, Severance Hospital, Yonsei University Health System, Seoul, South Korea